CLINICAL TRIAL: NCT04750642
Title: Cochlear Implant With Dexamethasone Eluting Electrode Array (The CI-DEX Study): Pivotal Study
Brief Title: Cochlear Implant With Dexamethasone Eluting Electrode Array
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: NAMSA (Other); Avania (Industry); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLTD5759
Record Dates: First submitted 2021-01-31; First posted 2021-02-11 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Sensorineural Hearing Loss; Bilateral Hearing Loss
Keywords: Cochlear Implant; Dexamethasone; Bilateral Hearing Loss; Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CI632D Investigational Medical Device (IMD) (Experimental)
  Interventions: Device: CI632D
- CI632 Comparator Device (Active Comparator)
  Interventions: Device: CI632

INTERVENTIONS:
Device: CI632D — CI632 cochlear implant with Slim Modiolar electrode including dexamethasone in the electrode within wells (CI632D)
  Arms: CI632D Investigational Medical Device (IMD)
Device: CI632 — CI632 cochlear implant with Slim Modiolar electrode with market approval and does not include dexamethasone
  Arms: CI632 Comparator Device

SUMMARY:
An evaluation of Cochlear's cochlear implant electrode array which passively elutes dexamethasone for a defined period of time to help reduce inflammatory responses.

DETAILED DESCRIPTION:
The primary objectives of the pivotal evaluation is to show the efficacy of the dexamethasone eluting electrode through reduction in electrode impedances as compared to a standard electrode and the improvement of speech recognition from preoperative baseline. The secondary objectives are to assess the benefit-risk balance of a dexamethasone eluting electrode as similar to a standard electrode by comparison of adverse events and speech outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Post-lingual, bilateral, moderate (≥ 40 dB HL) to profound sensorineural hearing loss at 250, 500and 1000 Hz and profound high-frequency hearing loss, defined by a pure-tone average (PTA) threshold, 2000 through 8000 Hz, ≥ 90 dB HL.
* 18 years or older at time of consent.

Exclusion Criteria:

* Abnormal cochlear and middle ear anatomy
* History with cochlear implant surgery
* Allergy to dexamethasone
* Women who are pregnant or plan to become pregnant
* Unable/unwilling to comply to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Parkinson, Study Director — Cochlear
Locations (8):
- United States (4):
  - Rocky Mountain Ear Centre, Englewood, Colorado
  - University of Iowa, Iowa City, Iowa
  - New York Eye & Ear infirmary of Mt. Sinai, New York, New York
  - NYU Langone Medical Center, New York, New York
- Australia (3):
  - Fiona Stanley Hospital, Murdoch, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
- Gilles Hospital, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Device
Started (Forty-two participants were enrolled in the study. Ten out of the 42 participants failed screening, and three subjects were eligible but withdrew prior to randomization with the decision to cease enrolment. Twenty-nine participants were randomized into the two groups (CI632D and CI632).) | 14 | 15
Completed | 13 | 13
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Device | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (8.5) | 66.3 (17.1) | 68.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 6 | 8 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Croatian | 1 | 0 | 1
  French Indian | 0 | 1 | 1
  Maori/European | 1 | 0 | 1
  White | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 1 | 2
  United States | 11 | 11 | 22
  Australia | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Monopolar (MP1+2) Impedance Measurement (kOhms) Between Randomization Groups at 6 Months Postoperative
Description: The impedance was measured across the active electrodes of the cochlear implant for each participant. Reduced impedances indicate less fibrotic obstruction caused by trauma associated with the electrode insertion.
Time Frame: Six months postoperative
Population: All implanted group. Thirteen participants in each arm completed the study. However, one participant from each arm did not complete the 6 month evaluation, which was the time frame for this outcome measure. Hence, the number of participants analyzed in each arm was 12.
Measure: Mean (Standard Deviation); unit: kOhms
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Device
Number analyzed (Participants) | 12 | 12
kOhms | 3.99 (0.54) | 8.66 (1.45)

2. Primary Outcome: Change in Speech Perception Performance (Pre-recorded CNC Words in Quiet in Sound Booth Testing) Compared to Pre-operative Baseline Measured at 6 Months Postoperative With CI632D
Description: Scores on the CNC Words in Quiet test were expressed as a percentage of words repeated correctly by the participant in a sound booth. A higher score indicates better speech perception performance. This outcome measure included the CI632D group only.
Time Frame: Six months postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | CI632D Investigational Medical Device (IMD)
Number analyzed (Participants) | 12
percentage points | 39.5 (23.1)

3. Secondary Outcome: Comparison of Rate and Type of Device Related Adverse Events Between Randomization Groups
Description: Adverse events were recorded from baseline to 12 months postoperative.
Time Frame: Twelve months postoperative
Population: Intent-to-treat group at 12 months. This is the number of participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Device
Number analyzed (Participants) | 14 | 15
Participants
  No adverse events | 2 | 3
  One or more AEs | 12 | 12
  One or more related (possibly, probably, definitely) AEs | 8 | 5
  Procedure related | 7 | 4
  Device related | 5 | 3
  Study drug related | 1 | 2
  One or more unanticipated adverse device effects (ADEs) | 0 | 0
  One or more serious AEs | 3 | 2
  One or more serious ADEs (SADEs) | 1 | 0
  One or more serious unanticipated ADEs (USADEs) | 0 | 0
  Discontinuation due to an AE | 1 | 0

4. Secondary Outcome: Comparison of Speech Perception Performance (Pre-recorded CNC Words in Quiet in Sound Booth Testing) Between the Randomization Groups at Six Months Postoperative
Description: Scores on the CNC Words in Quiet test were expressed as a percentage of words repeated correctly by the participant in a sound booth. A higher score indicates better speech perception performance.
Time Frame: Six months postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage points
Groups:
- CI632 Comparator Arm: Standard CI632 device
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Arm
Number analyzed (Participants) | 12 | 12
percentage points | 57.8 (17.6) | 68.0 (23.9)

5. Secondary Outcome: Comparison of Speech Perception Performance (AzBio Sentences in Quiet in Sound Booth Testing) Between Randomization Groups at Six Months Postoperative
Description: Scores from the AzBio Sentences in Quiet test were expressed as a percentage of words repeated correctly by the participant in a sound booth. A higher score indicates better speech perception performance.
Time Frame: Six months postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Arm
Number analyzed (Participants) | 12 | 12
percentage correct | 46.1 (35.3) | 55.3 (31.8)

ADVERSE EVENTS:
Time Frame: Baseline to 12 months postoperative
Arm/Group | CI632D Investigational Medical Device (IMD) | CI632 Comparator Arm
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/14 | 2/15
Other Adverse Events (participants affected / at risk) | 9/14 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CI632D Investigational Medical Device (IMD) (N=14) | CI632 Comparator Arm (N=15)
Reimplantation due to electrode tip fold over (Surgical and medical procedures) | 1 | 0 — The event was classified as serious because rehospitalization was required to replace the implant
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CI632D Investigational Medical Device (IMD) (N=14) | CI632 Comparator Arm (N=15)
Tinnitus (Ear and labyrinth disorders) | 2 | 6
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypoglycemia (Endocrine disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
(Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Discomfort (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Hypertension (General disorders) | 0 | 1
Wound dehiscence (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0
Viral infection (Infections and infestations) | 1 | 3
Bruise (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance problems (Nervous system disorders) | 3 | 1
Cognitive changes (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 9 | 6
Numbness (Nervous system disorders) | 0 | 1
Undesired nerve stimulation (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Abscess (Skin and subcutaneous tissue disorders) | 0 | 1
Itching sensation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Implant pain (Surgical and medical procedures) | 2 | 1
Inadequate pain relief (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
Early study termination leading to small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT04750642/Prot_001.pdf